CLINICAL TRIAL: NCT00840073
Title: A Single-Dose, Comparative Bioavailability Study of Two Formulations of Trandolapril 4 mg Tablets Under Fed Conditions.
Brief Title: Trandolapril 4 mg Tablet Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2004-842
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — trandolapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trandolapril (Experimental): Trandolapril 4 mg Tablet (test) dosed in first period followed by Mavik® 4 mg Tablet (reference) dosed in second period
  Interventions: Drug: Trandolapril 4 mg Tablets
- Mavik® (Active Comparator): Mavik® 4 mg Tablet (reference) dosed in first period followed by Trandolapril 4 mg Tablet (test) dosed in second period
  Interventions: Drug: Mavik® 4 mg Tablets

INTERVENTIONS:
Drug: Trandolapril 4 mg Tablets — 1 x 4 mg, single-dose fed
  Arms: Trandolapril
Drug: Mavik® 4 mg Tablets — 1 x 4 mg, single-dose fed
  Arms: Mavik®

SUMMARY:
The objective of this study is to evaluate the comparative bioavailability between trandolapril 4 mg tablets (test) and Mavik® 4 mg Tablets (reference) after a single-dose in healthy subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects, 18 years of age or older.
* BMI greater than or equal to 19 and less than or equal to 30.
* Negative for HIV, Hepatitis B surface antigen and Hepatitis C antibody, urine drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone), urine cotinine test, serum HCG consistent with pregnancy (females only).
* No significant diseases or clinically significant findings in a physical examination.
* No clinically significant abnormal laboratory values.
* No clinically significant findings in the 12-lead electrocardiogram (ECG).
* Blood pressure over 90/60 mmHg and less than 140/90 mmHg.
* Be informed of the nature of the study and given written consent prior to receiving any study procedure.
* Females who are surgically sterile for at least six months or postmenopausal for at least one year, or who will avoid pregnancy prior to the study, during the study and up to one month after the end of the study.
* Females who participate in this study are not pregnant and/or non-lactating.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition.
* Known history of food allergies, or any condition know to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Known or suspected carcinoma.
* Presence or history of angioedema.
* Known history or presence of hypersensitivity or idiosyncratic reaction to trandolapril and/or any other drug substances with similar activity; alcoholism within the last 12 months; drug dependence and/or substance abuse; use of tobacco or nicotine-containing products, within the last 6 months.
* Any clinically significant illness or surgery within 4 weeks prior to drug administration.
* On a special diet within 4 weeks prior to drug administration (e.g. liquid, protein, raw food diet).
* Participated in another clinical trial or received an investigational product within 30 days prior to drug administration.
* Donated up to 250 mL of blood within the previous 30 days OR donated from 251 to 500 mL of blood in the previous 45 days OR donated more than 500 mL of blood in the previous 56 days (based on the Canadian Blood Services guideline for blood donation).
* Use of any prescription medication within 14 days prior to period 1 dosing. Use of any over the counter (OTC) medication within 7 days prior to period 1 dosing (except spermicidal/barrier contraceptive products).
* Use of any drug known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoine, glucocorticoids, omeprazole; examples of inhibitors: antidepressant (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to period 1 dosing.
* Females taking oral or transdermal hormonal contraceptives within 30 days preceding period 1 dosing OR Females having taken implanted or injected hormonal contraceptives (Depo-Provera) within one year prior to period 1 dosing.
* Difficulty fasting or consuming the standard meals.
* Do not tolerate venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-10; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, M.D., Ph. D., Principal Investigator — Pharma Medica
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Trandolapril (Test) First: Trandolapril 4 mg Tablet (test) dosed in first period followed by Mavik® 4 mg Tablet (reference) dosed in second period
- Mavik® (Reference) First: Mavik® 4 mg Tablet (reference) dosed in first period followed by Trandolapril 4 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Trandolapril (Test) First | Mavik® (Reference) First
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Trandolapril (Test) First | Mavik® (Reference) First
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Missed 72 hour blood draw | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trandolapril (Test) First | Mavik® (Reference) First | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 17 | 18 | 35
  Black | 6 | 4 | 10
  Asian | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis. Data from two subjects who did not complete was also included in statistical analysis since the 72 hour blood draw that was missed does not affect the results for Trandolapril.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Trandolapril: Trandolapril 4 mg Tablet (test) dosed in either period
- Mavik®: Mavik® 4 mg Tablet (reference) dosed in either period
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 50 | 50
ng/mL | 5.2604 (3.8238) | 5.4938 (3.7393)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 96.00, 90% CI [85.13 to 108.27] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis. Not all data from completed subjects could be used to determine AUC0-inf.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 20 | 22
ng*h/mL | 7.0104 (1.9298) | 7.9967 (2.8867)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 103.81, 90% CI [96.72 to 111.41] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 50 | 50
ng*h/mL | 6.9056 (2.7329) | 6.7143 (2.4740)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 102.37, 90% CI [97.34 to 107.65] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

4. Secondary Outcome: Cmax - Trandolaprilat
Description: Informational Purposes Only
Time Frame: Blood samples collected over 72 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 50 | 50
ng/mL | 6.9610 (2.5672) | 6.6815 (2.4413)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 103.76, 90% CI [100.08 to 107.57] — Informational Purposes Only

5. Secondary Outcome: AUC0-72 - Trandolaprilat
Description: Informational Purposes Only
Time Frame: Blood samples collected over 72 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 50 | 50
ng*h/mL | 127.6059 (23.9616) | 123.4560 (22.6436)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Least Squares Means = 103.34, 90% CI [100.84 to 105.92] — Informational Purposes Only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.